CLINICAL TRIAL: NCT01031810
Title: Developing a Biomarker to Predict Response in Treatment Resistant Depression
Brief Title: PET Biomarkers in Treatment Resistant Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Needed PET facility closed
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6025; RC1MH088405-01 (NIH)
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: Treatment Resistant depression; Major Depression; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Tranylcypromine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tranylcypromine (Other): patients will receive treatment with tranylcypromine
  Interventions: Drug: tranylcypromine

INTERVENTIONS:
Drug: tranylcypromine — MAO-Inhibitor 60mg-120mg
  Other Names: Parnate

SUMMARY:
The primary objectives of the study are to test whether brain Mono Amine Oxidase-A (MAO-A) levels are elevated in patients with treatment-resistant major depression, and to explore whether MAO-A brain levels predict treatment outcome with Mono Amine Oxidase Inhibitor (MAOI) medication in this population.

DETAILED DESCRIPTION:
While Major Depressive Disorder (MDD) is prevalent and disabling, compelling recent data from the Sequenced Treatment Alternatives to Relieve Depression (STAR*D) study indicate that only about half of patients attain remission from MDD, even after multiple antidepressant medication trials. Further, no biomarker has been validated which can select an effective treatment for such patients, presenting critical unmet intellectual and clinical challenges. The recent landmark finding of an markedly elevated level of monoamine oxidase A (MAO-A) in the brains of depressed patients with MDD compared to controls, using positron emission tomography (PET) with a positron-emitting carbon isotope, (carbon 11 [11C]) labeled monoamine oxidase inhibitor (MAOI), has provided an unparalleled opportunity to address these challenges. It has long been known that MAOIs are effective for some patients with treatment-resistant MDD, although their side effect profile makes them highly unacceptable both to patients and physicians, severely curtailing their utility.

This study seeks to: 1) replicate this study using PET scans in 20 subjects with MDD but extending it to patients with treatment-resistant depression (TRD). (Results from these participants with be compared to those from 10 non-depressed controls; 2) explore the correlation of the brain MAO-A level biomarker to treatment outcome by treating the 20 PET-imaged TRD patients with an MAOI, hypothesizing that their MAOI response will be related to their level of MAO-A. Brain MAO-A is an ideal candidate biomarker for this study since it appears to be significantly abnormally elevated in MDD, yet it has a broad range of values even among depressed patients. Most importantly, the MAO-A biomarker is known to be the single pharmacologic target of the treatment, making it appear likely that outcome with MAOI treatment will be related to MAO-A.

ELIGIBILITY:
INCLUSION:

1. Primary diagnosis of Major Depressive Disorder
2. Subjects aged 18-65
3. Depressed subjects must have Treatment-Resistant Depression (TRD) two previous adequate antidepressant treatment trial failures within the current depressive episode from different classes
4. Minimum baseline Montgomery Asberg Depression Rating Scale (MADRS) score of 22
5. Signs informed consent form
6. Subjects must be willing to be have a PET scan
7. Subjects must be antidepressant medication free for 3 weeks prior to PET scan

EXCLUSION

1. Significant past or present neurological disorder, including seizures, stroke, or head trauma
2. History of bipolar disorder, psychosis, schizoaffective disorder, or schizophrenia
3. Moderate or high level of suicide risk, as determined by a score of 3 or 4 on item 3 of the HAM-D scale. Also excluded will be those who present a significant suicide risk by history or current psychiatrist's assessment.
4. Personality disorder which might interfere with compliance or increase suicide risk
5. Alcohol or drug abuse or dependence in the past year; history of lifetime IV drug use or use of methylene diamine methamphetamine (MDMA or "ecstasy") more than twice
6. Current thyroid dysfunction (past or currently treated dysfunction is acceptable)
7. Clinically significant or unstable medical conditions or laboratory abnormalities, including hypertension (repeated BP > 140 systolic, > 90 diastolic)
8. Intake of investigational (unapproved) drug in the past 3 months
9. Electroconvulsive therapy (ECT) in three months prior to screening
10. Use of Vagal Nerve Stimulation (VNS)
11. Positive drug of abuse screen
12. Anticoagulant treatment which cannot be discontinued for 10 days prior to PET scanning
13. Pregnancy, currently lactating; planning to conceive during the course of study participation or abortion in the past two months.
14. Dementia (clinical and neurocognitive criteria)
15. Claustrophobia of a severity which would not permit the participant to undergo an MRI or a PET scan
16. Recent (< 7 days) consumption of Ayahuasca Tea or other South American non-standard decoction.
17. Presence of metallic devices, implants and other contraindications to scanning
18. Current, past or anticipated exposure to radiation, that may include being badged for radiation exposure in the workplace or participation in nuclear medicine research protocols
19. Smokers (use of tobacco products in the previous 3 months)
20. Potential participants having taken an antidepressant medication in the last 3 weeks. Participants otherwise eligible may elect to discontinue medication which has not been significantly helpful according to their report, their current psychiatrist's report (if available), and the evaluating psychiatrist. No patient will be asked to discontinue an effective antidepressant medication to participate.
21. History of previous MAO-I treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, MD, Principal Investigator — New York State Psychiatric Institute, Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Depression Evaluation Service website — http://depression-nyc.org
- See also: New York State Psychiatric Institute official website — http://nyspi.org/
- See also: Columbia University Psychiatry website — http://www.cumc.columbia.edu/dept/pi/

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranylcypromine: Patients will receive treatment with tranylcypromine tablets taken orally on a twice daily schedule. Dosage was initially 10 mg daily and was increased weekly up to 120 mg daily.
Period: Overall Study
Arm/Group | Tranylcypromine
Started | 13
Completed | 9
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale Scores 17 at Baseline
Description: HAM-D is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. Each item on the questionnaire is scored on a 3 or 5 point scale, depending on the item, and the total score is compared to the corresponding descriptor.
  Scale range (0-52):
  A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression, and are usually required for entry into a clinical trial.
Time Frame: Week 00 (baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tranylcypromine: patients will receive treatment with tranylcypromine Baseline Hamd17
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 9
units on a scale | 23.2 (5.8)
Statistical Analysis 1: Comparison: Tranylcypromine; Compare the mean differences between baseline (week00) and week12 hamd17 summary scores; Test type: Superiority or Other; p = 0.012, paired t-test 2 sided; Mean Difference (Final Values) = 11.56, 95% CI 2-sided [3.25 to 19.86], Standard Deviation 10.81

2. Secondary Outcome: Quick Inventory of Depression- Self Report 16
Description: Quick Inventory of Depression- Self Report assesses 16 depressive symptoms experienced in the past week, based on self-rating, measured at study exit visit
  Scale range (0-27):
  Each of the four possible answers to each quiz is given an ascending numerical value from 0 to 3, and the total test score is the sum of the following: The highest number from questions 1-4 The number from question 5 The highest number from questions 6-9 The total of each question from 10-14 The highest number from questions 15-16
  Total score interpretation: 0-5 no depression, 6-10 mild depression, 11-15 moderate depression, 16-20 severe depression, 20 and above very severe depression
Time Frame: Weeks 00
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tranylcypromine: patients will receive treatment with tranylcypromine
  tranylcypromine: monoamine oxidase inhibitor (MAOI) 60mg-120mg
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 9
units on a scale | 17.78 (3.03)

3. Secondary Outcome: Quick Inventory of Depression- Self Report 16
Description: as for outcome 2
Time Frame: Week 04
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 9
units on a scale | 13.0 (6.27)

4. Secondary Outcome: Quick Inventory of Depression- Self Report 16
Description: as for outcome 2
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 9
units on a scale | 10.38 (5.04)

5. Secondary Outcome: Quick Inventory of Depression- Self Report 16
Description: as for outcome 2
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 9
units on a scale | 9.89 (5.23)

6. Primary Outcome: Hamilton Depression Rating Scale Scores 17 at week12
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 9
Score on a scale | 11.67 (6.29)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected weekly from baseline(week 00) to week 16.
Arm/Group | Tranylcypromine
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranylcypromine (N=9)
Constipation (Gastrointestinal disorders) | 4 (4)
Dizziness (General disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes